CLINICAL TRIAL: NCT04793386
Title: Usefulness of the Evaluation of the Return of Spontaneous Circulation(ROSC) With Carotid Ultrasound During Cardiopulmonary Resuscitation(CPR)
Brief Title: Usefulness of the Evaluation of the ROSC With Carotid Ultrasound During CPR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-11-116
Record Dates: First submitted 2021-02-14; First posted 2021-03-11 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-02

CONDITIONS: Cardiopulmonary Arrest
MeSH Terms: conditions — Heart Arrest | interventions — Ultrasonography, Carotid Arteries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Carotid ultrasound (Experimental): When stopping chest compressions to check manual palpation every 2 minutes, an ultrasound scan of the carotid artery is performed. Whether or not return of spontaneous circulation is determined based on the compressibility and pulsatility of the carotid artery, and the time taken from the start of the ultrasound scan to the determination is recorded.
  Interventions: Diagnostic Test: carotid ultrasound

INTERVENTIONS:
Diagnostic Test: carotid ultrasound — Every time checking pulse, evaluate the carotid artery compressibility and pulsatility by ultrasound

SUMMARY:
The current cardiopulmonary resuscitation(CPR) guidelines recommend that the heart rhythm be checked every two minutes during CPR for cardiac arrest patients. Also it is very important to stop compressing the chest in less than 10 seconds when checking heart rhythm and pulse.

However, manual palpation, which is used as a standard for return of spontaneous circulation(ROSC), has been reported that the accuracy is not high in several studies. It is quite often necessary to perform pulse palpation for longer than the 10 second recommended by the guidelines to make a judgment.

Recently, a case study was published in which the presence of spontaneous circulation was confirmed by evaluating the carotid artery compressibility and pulsatility with an ultrasound probe when checking the rhythm of cardiac arrest patients. However, there has been no clinical study on actual cardiac arrest patients.

DETAILED DESCRIPTION:
The current cardiopulmonary resuscitation(CPR) guidelines recommend that the heart rhythm be checked every two minutes during CPR for cardiac arrest patients. Also it is very important to stop compressing the chest in less than 10 seconds when checking heart rhythm and pulse.

However, manual palpation, which is used as a standard for return of spontaneous circulation(ROSC), has been reported that the accuracy is not high in several studies. It is quite often necessary to perform pulse palpation for longer than the 10 second recommended by the guidelines to make a judgment.

Ultrasound is a key technique that guides to discern and treat causes of cardiac arrest patients. Recently, a case study was published in which the presence of spontaneous circulation was confirmed by evaluating the carotid artery compressibility and pulsatility with an ultrasound probe when checking the rhythm of cardiac arrest patients.

However, this is just a case study. There has been no clinical study on actual cardiac arrest patients whether it is possible to accurately determine the ROSC by evaluating the carotid artery compressibility and pulsatility by ultrasound. Also there has been no clinical studies on actual cardiac arrest patients comparing the time taken to evaluate the ROSC of carotid ultrasound and manual palpation.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent CPR among cardiac arrest patients 18 years of age or older who visit the emergency room
* Patients who applied carotid ultrasound to determine the presence of carotid artery compression and pulse

Exclusion Criteria:

* Patients who have stated their intention to do not resuscitation for future treatment (including cardiopulmonary resuscitation)
* Patients who have difficulty applying carotid ultrasound due to head and neck trauma
* Patients who have difficulty applying carotid ultrasound due to deformed neck structure by surgery or head and neck cancer
* Return of spontaneous circulation before ultrasound application
* Patients who could not evaluate carotid artery compressibility and pulsatility by ultrasound

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Time spent assessing | Procedure (during chest compression)
  Time spent assessing return of spontaneous circulation using two methods (manual pulse palpation and carotid ultrasound)

SECONDARY OUTCOMES:
Agreement of return of spontaneous circulation | Procedure (during chest compression)
  Compare the agreement between two methods (manual pulse palpation and carotid ultrasound) for evaluation of return of spontaneous circulation (ROSC).
  The gold standard is arterial blood pressure by arterial catheter. The ROSC is judged when pulsation is detected by manual palpation. The ROSC is judged when carotid artery is not totally compressed or has pulsatility by carotid artery ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Hee Yoon, Professor, Study Chair — Samsung medical center, Emergency department
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No